CLINICAL TRIAL: NCT00815802
Title: Detection of Human Cytomegalovirus in the Saliva of 3 Month to 6 Year-Old Children in Day Care Centers : a Pilot Study.
Brief Title: Detection of Human Cytomegalovirus in the Saliva
Acronym: FcrèchMV
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Other Study IDs: I07017
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Cytomegalovirus
Keywords: Children in day care centers; cytomegalovirus excretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Direct DNA amplification, viral isolation and specific antibody measurement in saliva

1. From children in day care centers (samples collection will take place during a single week)
2. From children coming at the emergency department of our hospital during a three months period.

Sample collection will be done by the pediatrician the nurse, or one of the authorized investigators of the study.

DETAILED DESCRIPTION:
Salivary collection kit. Collection of salivary at the internal face of the mooth. 3 swab for DNA research, 1 for antibodies research and 1 for virus isolation by cell growth.

ELIGIBILITY:
Inclusion Criteria:

* parents consent
* child aged from 3months to 6 years
* child in day care centers or emergency department

Exclusion Criteria:

* Refuse of participation

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: child aged from 3 month to 6 years in day care centers or in emergency department.
Sampling Method: Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2007-07

PRIMARY OUTCOMES:
One week trial of saliva sampling for cytomegalovirus detection in day-care centers.

SECONDARY OUTCOMES:
Percentage of chidrens with CMV excretion among those coming at the Emergency department of Limoges teacher Hospital (CHU). Validation of the process from samples collection to interpretation of results

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ALAIN, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Bactériologie-Virologie, Limoges, France